CLINICAL TRIAL: NCT02254577
Title: A Randomized, Three-armed, Non-Inferiority Study of Vaginal Progesterone (Endometrin®) Compared to Intramuscular Progesterone in Oil (PIO) in Infertile Subjects Undergoing Frozen Embryo Transfer (FET)
Brief Title: Vaginal Compared to Intramuscular Progesterone for Frozen Embryo Transfer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shady Grove Fertility Reproductive Science Center (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0028; SUSTAIN (Other: ShadyGroveFRSC)
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Infertility
Keywords: Infertility; Progesterone; ART; IVF; FET; FBT; Frozen Embryo Transfer
MeSH Terms: conditions — Infertility | interventions — Progesterone; Oils; Sesame Oil; Pemoline; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endometrin® plus Progesterone in Oil (PIO) (Experimental): Subjects in all arms will undergo the standard monitoring appointments and therapies involved in a frozen embryo transfer cycle. Patients randomized to the Endometrin® plus PIO arm will take progesterone as 2 100mg tablets of Endometrin® inserted vaginally twice daily. In addition, on the first day of Endometrin® therapy, patients randomized to this arm will take a 50mg intramuscular injection (1mL) of PIO and will repeat this injection every third day. Patients in this arm will undergo Frozen Embryo Transfer on the fifth day of Endometrin® therapy.
  Interventions: Drug: Endometrin® plus Progesterone in Oil (PIO)
- Progesterone in Oil (PIO) Alone (Active Comparator): Subjects in all arms will undergo the standard monitoring appointments and therapies involved in a frozen embryo transfer cycle. Patients randomized to the PIO Only arm will take progesterone as a daily 50mg intramuscular injection (1mL) of PIO and will undergo Frozen Embryo Transfer on the sixth day of taking this medication.
  Interventions: Drug: Progesterone in Oil (PIO) Only

INTERVENTIONS:
Drug: Endometrin® plus Progesterone in Oil (PIO)
  Other Names: Vaginal Micronized Progesterone Tablet; Progesterone in Sesame Oil Injection
  Arms: Endometrin® plus Progesterone in Oil (PIO)
Drug: Progesterone in Oil (PIO) Only
  Other Names: Progesterone in Sesame Oil Injection
  Arms: Progesterone in Oil (PIO) Alone

SUMMARY:
To determine whether the of vaginal progesterone replacement for frozen embryo transfer results in equivalent live birth rates to intramuscular injection progesterone replacement.

DETAILED DESCRIPTION:
The purpose of this ongoing study is to look at whether Endometrin® (vaginal micronized progesterone tablets) supplemented by intramuscular injection of progesterone in oil (PIO) work as well as PIO alone for women undergoing transfer of frozen-thawed blastocyst(s). Another goal of the study is to determine whether patients prefer Endometrin or PIO. Endometrin® has been approved by the United States Food and Drug Administration, or FDA, "to support embryo implantation and early pregnancy by supplementation of corpus luteal function as part of an Assisted Reproductive Technology (ART) treatment program for infertile women." (FDA New Drug Approval Letter, Endometrin®, 2007). The use of Endometrin® (vaginal micronized progesterone tablets) in this study is investigational. An investigational use is one that is not approved by the U.S. Food and Drug Administration (FDA).

Approximately 1170 women between the ages of 18-48 who are having difficulty becoming pregnant and wish to undergo frozen embryo transfer will be asked to participate. The participants will be recruited from among patients of Shady Grove Fertility.

One-half of the participants who qualify and wish to take part in the ongoing study will be randomized (assigned by chance, like the flip of a coin) to receive Endometrin® and an intramuscular injection of PIO every third day. One-half will be randomized to receive an intramuscular injection of PIO every day. This study is a type of study called an "open label," assessor-blind study. This means that you and your doctor will know which treatment you are assigned and receive; however, the person analyzing the information obtained from the study will not know which patients received which study treatments.

Patients enrolling in the study will receive the medications for their frozen embryo transfer cycle free of charge.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Female age between 18 and 48 years
3. Having available blastocyst(s) frozen by vitrification method at our center (Shady Grove Fertility).
4. Standard eligibility criteria to undergo frozen blastocyst transfer at Shady Grove Fertility.

Exclusion Criteria:

1. Requires fresh embryos or surrogate carrier
2. Embryos from frozen oocytes and embryos frozen more than once
3. Any embryo cryopreserved by slow freeze method and/or prior to blastocyst stage
4. Presence of any clinically relevant systemic disease contraindicated for ART
5. History of more than 3 failed cycles in previous ART attempts and/or more than 3 recurrent pregnancy losses after ET
6. Surgical or medical condition or requirement for medication, which may interfere with absorption, distribution, metabolism, or excretion of the drugs to be used
7. Subjects with a body mass index (BMI) of <18 or >38 kg/m2 at screening
8. Current or recent substance abuse, including alcohol and tobacco. (Note: Subjects who stopped tobacco usage at least 3 months prior to screening visit will be allowed)
9. Currently breast feeding, pregnant, or having (a) contraindication(s) to pregnancy
10. Refusal or inability to comply with the requirements of the protocol for any reason, including scheduled clinic visits and laboratory tests
11. Trophectoderm or blastomere biopsy of the blastocyst(s) to be transferred.
12. Documented intolerance or allergy to any of the medications used, including the study medication
13. Participation in any experimental drug study within 60 days prior to screening
14. If a subject undergoes more than two frozen blastocyst transfers meeting study criteria, she will only be eligible to enroll in the study for two of these.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1139 (Actual)
Dates: Start 2014-10; Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Live Birth | ~40 weeks post Frozen Embryo Transfer
  Live born infant at 23 weeks' estimated gestational age or greater.

SECONDARY OUTCOMES:
Ongoing Implantation Rate | 7-8 weeks after embryo transfer
  maximum # fetal heartbeats divided by total number of embryos transferred
Implantation rate | 5-6 weeks post embryo transfer
  Maximum number of gestational sacs, divided by total number of embryos transferred
Biochemical pregnancy | ~10 days following embryo transfer
  detection of beta hCG (pregnancy hormone) above 5 IU/L
Clinical pregnancy | 5-6 weeks following embryo transfer
  Presence of gestational sac(s) at 5-6 weeks post ET
Serum progesterone level | ~10 days following embryo transfer
  blood draw
Patient satisfaction with Endometrin® vs. intramuscular progesterone in oil | between 0 and 10 days following embryo transfer
  As assessed by brief, optional online survey

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Shady Grove Fertility Center, Washington D.C., District of Columbia
  - Shady Grove Fertility Center, Annapolis, Maryland
  - Shady Grove Fertility Center, Baltimore, Maryland
  - Shady Grove Fertility Center, Bel Air, Maryland
  - Shady Grove Fertility Center, Columbia, Maryland
  - Shady Grove Fertility Center, Frederick, Maryland
  - Shady Grove Fertility Center, Rockville, Maryland
  - Shady Grove Fertility Center, Towson, Maryland
  - Shady Grove Fertility, Camp Hill, Pennsylvania
  - Shady Grove Fertility Center, Chesterbrook, Pennsylvania
  - Shady Grove Fertility Center, Annandale, Virginia
  - Shady Grove Fertility Center, Leesburg, Virginia
  - Shady Grove Fertility Center, Woodbridge, Virginia

REFERENCES:
- [Background] Shapiro DB, Pappadakis JA, Ellsworth NM, Hait HI, Nagy ZP. Progesterone replacement with vaginal gel versus i.m. injection: cycle and pregnancy outcomes in IVF patients receiving vitrified blastocysts. Hum Reprod. 2014 Aug;29(8):1706-11. doi: 10.1093/humrep/deu121. Epub 2014 May 20. PMID 24847018
- [Background] Feinberg EC, Beltsos AN, Nicolaou E, Marut EL, Uhler ML. Endometrin as luteal phase support in assisted reproduction. Fertil Steril. 2013 Jan;99(1):174-178.e1. doi: 10.1016/j.fertnstert.2012.09.019. Epub 2012 Nov 6. PMID 23137759
- [Background] Paulson RJ, Collins MG, Yankov VI. Progesterone pharmacokinetics and pharmacodynamics with 3 dosages and 2 regimens of an effervescent micronized progesterone vaginal insert. J Clin Endocrinol Metab. 2014 Nov;99(11):4241-9. doi: 10.1210/jc.2013-3937. Epub 2014 Feb 25. PMID 24606090
- [Derived] Devine K, Richter KS, Jahandideh S, Widra EA, McKeeby JL. Intramuscular progesterone optimizes live birth from programmed frozen embryo transfer: a randomized clinical trial. Fertil Steril. 2021 Sep;116(3):633-643. doi: 10.1016/j.fertnstert.2021.04.013. Epub 2021 May 13. PMID 33992421
- [Derived] Devine K, Richter KS, Widra EA, McKeeby JL. Vitrified blastocyst transfer cycles with the use of only vaginal progesterone replacement with Endometrin have inferior ongoing pregnancy rates: results from the planned interim analysis of a three-arm randomized controlled noninferiority trial. Fertil Steril. 2018 Feb;109(2):266-275. doi: 10.1016/j.fertnstert.2017.11.004. Epub 2018 Jan 17. PMID 29338855